CLINICAL TRIAL: NCT03649334
Title: Analgesic Efficacy of Intra-muscular Ketamine-ketorolac Versus Fentanyl- Ketorolac for Children Undergoing Bone Marrow Biopsy and Aspiration
Brief Title: Ketamine-ketorolac Versus Fentanyl- Ketorolac I.M in Children During Bone Marrow Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R/18.06.213
Record Dates: First submitted 2018-08-18; First posted 2018-08-28 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Hematological Malignancy (Leukemia- Lymphoma)
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine-ketorolac (Other): The patient will receive ketamine in conjunction with intramuscular ketorolac
  Interventions: Drug: ketamine-ketorolac
- fentanyl- ketorolac (Other): The patient will receive fentanyl in conjunction with intramuscular ketorolac
  Interventions: Drug: fentanyl- ketorolac

INTERVENTIONS:
Drug: ketamine-ketorolac — The patient will receive ketamine 0.5mg.kg-1 + ketorolac 1mk.kg-1 in 2 ml syringe intramuscularly.
  Arms: ketamine-ketorolac
Drug: fentanyl- ketorolac — The patient will receive fentanyl 1.5ug.kg-1 + ketorolac 1 mg.kg-1 in 2ml syringe intramuscularly
  Arms: fentanyl- ketorolac

SUMMARY:
investigators aim to compare between anaesthetic regimens that included dual-agent (fentanyl and ketorolac) or (ketamine and ketorolac) analgesic therapy

DETAILED DESCRIPTION:
regarding patient registry; a prior G power analysis was done. Based on the assumption that the pain score in intramuscular ketamine group will be similar to similar to those in previously published data; forty children would be required per group to detect a difference of 30% in CHEOPS pain scores with a power of 90% (α =0.05, β =0.1)

- Statistical analysis: Data will be analyzed through SPSS (Statistical Package for Social Sciences), program version 22. Distribution of data will be first tested by the Shapiro test. Data will be presented as the mean and standard deviation (SD), median and range or numbers and percentages. For normally distributed data, the unpaired t-test will be used to compare the mean values of both groups. For pain and emergence behaviour scores, Mann Whitney U test will be used. Fisher's exact test will be used for comparison of categorical data. The P value ≤ 0.05 will be considered as the level of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status II

Exclusion Criteria:

* Any known allergy to the studied drugs.
* congenital heart disease
* Any cardiac problems.
* Use of psychotropic medication
* mental retardation
* any organ dysfunction

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | for 60 minutes later admission to the post-anaesthesia care unit
  Postoperative pain will be assessed by the CHEOP scale (Children's Hospital of Eastern Ontario Pain Scale)The scale includes six entries with an appropriate point evaluation focused on the character of crying (1-3 points), facial expressions (0-2 points), verbal reaction (0-2 points), position of the body (1-2 points), touch (1-2 points), and position of the legs (1-2 points). Minimum score is 4 (no pain) and maximum is 13 (maximum pain). Grades are summed together. CHEOPS has a minimum possible score of 4 points (no pain) to a maximum of 13 points (the worst pain).
  When the postoperative pain score exceeded four, rescue analgesia was given with a 20mg/kg paracetamol suppository.

SECONDARY OUTCOMES:
Heart rate | at the baseline (after the induction of anesthesia and before administration of the drugs) then every 5min up to 20 minutes
  Heart rate (beat/minute) using ECG monitoring
systolic blood pressure | at the baseline (after the induction of anesthesia and before administration of the drugs) then every 5min up to 20 minutes
  systolic blood pressure (mmHg) using sphygmomanometer cuff
The time to the first demand for rescue analgesic | during first 24 hours postoperative
  The time to the first demand for rescue analgesic (minutes or hours)
total number of children who required postoperative pain medication | for 24 hours after surgery
emergence behavior | every 5 minutes during first 30 minutes of recovery
  -emergence behavior will be measured using Aono's four point scale : (1) Asleep; (2) Awake but calm; (3) Agitated but consolable; and (4) Severely agitated and difficult to console and the highest-recorded value was recorded during the Post anesthesia care unit stay. Lowest score is 1 and highest score is 4 The higher score indicates more emergence agitation. For purposes of analysis, grades 1 and 2 in the scale of behavior were considered no agitation and grades 3 and 4 were considered the presence of agitation.
nausea, vomiting | during first 24 hours postoperative
  Number of attacks of nausea and/or vomiting
respiratory difficulty | during first 24 hours postoperative
  signs of respiratory difficulty:
  1. Breathing rate. An increase in the number of breaths per minute (>35 breath/minute)
  2. Increased heart rate.
  3. Color changes. A bluish color seen around the mouth, on the inside of the lips, or on the fingernails
  4. Grunting. A grunting sound can be heard each time the person exhales.
  5. Nose flaring. The openings of the nose spreading open while breathing
  6. Retractions. The chest appears to sink in just below the neck and/or under the breastbone with each breath-
  7. Sweating. There may be increased sweat on the head, but the skin does not feel warm to

CONTACTS AND LOCATIONS:
Overall Officials: Enas A Abd el Motlb, MD, Study Chair — Assisitant Professor
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided